CLINICAL TRIAL: NCT03455361
Title: Clinical Osteointegration of Bone Level Implants With Conical Shape and Textured Surface With Low Primary Stability
Brief Title: Evaluation of Bone Level Around Stark Conical Screw Implants With V-Blast Surface
Acronym: STARKIMPLANT
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giulio Rasperini, Professor, University of Milan
Other Study IDs: StarkImplant
Record Dates: First submitted 2018-02-16; First posted 2018-03-06 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Dental Impaction
Keywords: implant stability, dental implants, primary stability
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stark Implant with low primary stability: Patient who had received bone level V-Blast implants with low primary stability.
  Interventions: Procedure: Stark Implant with low primary stability
- Stark Implant with primary stability: Patient who had received bone level V-Blast implants and achieved primary stability.
  Interventions: Procedure: Stark Implant with low primary stability

INTERVENTIONS:
Procedure: Stark Implant with low primary stability

SUMMARY:
Clinical evaluation of osteointegration of bone level implants (Stark conical screw implants, with V-Blast surface treatment), placed without sufficient primary stability.

DETAILED DESCRIPTION:
26 Implants were placed with a unique operative protocol in 4 private offices. A detailed informed consent was obtained from all patients. Surgical guides were used to achieve the idea implant position and axis.

Osteotomy drills were used in the sequence recommended by the implant manufacturer. Bone type was assessed by CT examinations using the classification proposed by Rebaudi.

All implants were tested by applying a lateral mild load with a probe in order to verify mobility immediately after placement.

Parameter used to assess a low primary stability were:

* insertion torque lower than 10 N / cm
* slight mobility of implant upon application of lateral load of 250 g After surgery, patients were instructed not to chew or to wear their removable dentures in the treated areas.

Follow-up post-operative visits were scheduled at 1 and 4 weeks. At 4-6 months after placement a periapical radiograph was taken, a torque/countertorque test of 30 Ncm was conducted and osteointegrated implants were restored. Patients were recalled, examined, and periapical radiographs were taken for a minimum of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patient who had received Stark bone level V-Blast implants in 4 private offices in Italy
* patient subscribed a detailed informed consent
* same surgical protocol was applied

Exclusion Criteria:

* patient without Stark implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the sample is composed by patients who had received Stark bone level V-Blast implants in 4 private offices in Italy. The same surgical protocol was used for all implants and a detailed informed consent was obtained from all patients, and included in their respective charts.
  For the study objective were enrolled patient who didn't achieved primary stability at the placement: 26 patient
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Osteointegration of V-Blast surface implant with low primary stability (<10 N/cm) after 4-6 months | 4 to 6 months
  After 4-6 months, implant without good primary stability were evaluatd. A periapical radiograph was taken, a torque/countertorque test of 30 Ncm was conducted and osteointegrated implants were restored.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Rasperini, Prof., Study Director — University of Milan